CLINICAL TRIAL: NCT05699941
Title: Efficacy of Ectoin® Inhalation Solution EIL07 as Supportive Treatment for Children and Adult With Mild to Moderate Asthma: a Post-Market Clinical Follow-up (PMCF) Study.
Brief Title: Multicentre Post-market Study of Ectoin® Inhalation Solution in Treatment of Asthma.
Acronym: EIL-AST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: btph-046-2021-EIL07
Record Dates: First submitted 2022-12-16; First posted 2023-01-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: Asthma in children; Asthma in adults
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Ectoin® Containing Inhalation Solution (EIL07) (Class-IIa MDD legacy medical device).
  Taken twice daily over the period of 3 weeks (treatment) Inhalation of the content of EIL07 single dose (2.5 mL) by using a mesh nebulizer device.
  Interventions: Device: Ectoin® Inhalation Solution

INTERVENTIONS:
Device: Ectoin® Inhalation Solution — Ectoin Inhalation Solution (Class-IIa Medical Device Directive (MDD) legacy medical device) is an isotonic, aqueous solution containing Ectoin 1.3 % and sea salt 0.6%. It is used for moistening the lung epithelium by the Ectoin hydro complex and supports the barrier function of the lung epithelium. The inhalation solution can be administered with jet, mesh, and ultrasound nebulizers.

SUMMARY:
The goal of this multi-centre, prospective, open-label, single-arm, post-market clinical follow-up study is to further strengthen the already existing clinical evidence for supportive treatment and symptoms alleviation in asthma by evaluating the clinical efficacy of Ectoin® Inhalation Solution in paediatric and adults patients with mild to moderate asthma.

DETAILED DESCRIPTION:
A multi-centre, prospective, open-label, post-market follow-up study according to Article 61 and Part-B Annex XIV Medical Device Regulation (MDR 2017/745) and conforming to International Organization for Standardization - Clinical investigation of medical devices for human subjects - Good clinical practice (ISO 14155:2020) requirements.

Study participation will be offered to patients with clinically diagnosed Asthma for which the Ectoin Inhalation Solution is indicated. The enrollment will be subject to an invitation by the investigators of the study sites among their paediatric and adult outpatients coming in for the consultation about asthma. Participation in the study will be, however, based on compliance with all the inclusion criteria and subsequent signed informed consent (ICF) including assent where applicable.

The duration of participation in the clinical study will be 42±2 days (6 weeks) from enrollment). The clinical investigation comprises 4 visits and 1 telephone call. During the study, Ectoin® Inhalation Solution will be used from Visit V2 onwards until V3 (3 weeks) according to the Instruction for Use (IFU). V3 marks the end-of-treatment. However, a follow-up will be conducted at V4 which will mark the end-of-study/ end-of-follow-up.

Visit 1: (D1): Screening, enrollment and training. The first visit will be used for acquiring ICF as per age requirements. Subsequently, the final screening assessment and training of PEF recording will be performed. Also, the Asthma Control Questionnaire (ACQ-7) to be filled out by enrolled patients on the day.

Minimum 3 days of training following V1 the morning Peak Expiratory Flow (mPEF) is to be measured in the morning upon awakening before taking any asthma controller/rescue medication. The evening Peak Expiratory Flow (ePEF) is to be measured at bedtime.

The baseline measurement will be represented by the mean of the 7 daily values recorded during the run-in period (week 1) and only after the aforesaid 3 days of training. The subject will measure mPEF and ePEF for at least 7 days and complete the patient diary as applicable (also mentioning asthma attack and exacerbation reporting, rescue medication if any). The V2 will be scheduled to respect this period of 7 days minimum for the baseline value of mPEF value.

Visit 2 (V2) - (Day 11-D13): EIL07 treatment start. Completion of Paediatric Asthma Quality of Life Questionnaire (PAQLQ), ACQ-7 and Asthma Quality of Life Questionnaire (AQLQ+12) questionnaires as applicable and Fractional exhaled Nitric Oxide (FeNO) assessment.

From V2 to V3 patients will have to comply with daily treatment with EIL07, twice daily measurements of peak inspiratory flow, and daily completion of the diary (asthma attack and asthma exacerbation reporting, rescue medication, adverse event/incident linked to EIL07 intake).

A Telephone call (D21±2) will be initiated by the study clinics for updates (if any) and to check patient compliance.

Visit 3 (V3) - (Day 33- D37): End of Treatment. The end-of-treatment assessment will be the mean of mPEF at end of week 4 along with a repeat of all on-site questionnaires and assessments performed at V2. Completion of PAQLQ, ACQ-7and AQLQ+12 questionnaires and FeNO assessment.

**However, no mean will be performed at the visit and will be calculated after the end-of-study to establish the secondary endpoint.

From V3 to V4 patients will have to continue to record twice-daily measurements of mPEF and ePEF as well as daily completion of the diary (asthma attack and asthma exacerbation reporting, rescue medication if any)

Visit 4 (V4) - (Day 40- Day 45): End of study/end of follow-up. As a follow-up, all applicable PEFs will be repeated/recorded. Completion of ACQ-7 questionnaire and FeNO assessment.

The primary endpoint is the change of the mPEF from baseline to the end-of-treatment period (in 3 weeks' time). The Peak Expiratory Flow (applicable for both mPEF and ePEF) is defined as the maximum speed of expiration as measured with the Smart Peakflow (best of 3 measurements)

Secondary Endpoints:

* Change in weekly mean evening Peak Expiratory Flow (ePEF).
* Change in weekly mean morning Peak Expiratory Flow (mPEF).
* Evolution of the mean number of days with rescue medication intakes.
* Change of quality of life questionnaires, Paediatric Asthma Quality of Life Questionnaire (PAQLQ) score is applicable for children up to 12 years and Asthma Quality of Life Questionnaire (AQLQ+12) is applicable for patients aged 12-years and older
* Change of asthma control questionnaire (ACQ-7)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged≥ 6 years to 60 (included)
2. A documented clinical history of asthma for a period of at least 6 months
3. Baseline mild to moderate uncontrolled asthma, defined as meeting at least one of the following:

   1. Forced Expiratory Volume in 1 Second (FEV1): 60%<FEV1 <95% predicted
   2. Asthma Control Questionnaire (ACQ-7): Score ≥1.5
4. In case of routine treatment with Inhaled Corticosteroids (ICS), maintenance therapy for 8 weeks or longer (stable dose ≥4 weeks before screening)
5. Patient who qualifies for EIL07 treatment according to the approved indication and in physician's opinion the participant will benefit from this treatment.
6. Able to use the Smart Peakflow meter (with the help of a caregiver in case of minors, if needed)
7. Signed informed consent from legally designated representatives (for minors) / adult patients
8. Signed assent from minors if applicable
9. Willingness of the participants to actively participate in the study and to come to the scheduled visits.

   Exclusion Criteria:
10. Treatment with Ectoin® for respiratory conditions (in past 8 weeks)
11. Pregnant or breastfeeding women
12. Participation in any other clinical study within the last 4 weeks prior to screening.
13. Experienced a respiratory tract infection in the 4 weeks prior to Visit 1.
14. Experienced an acute asthma exacerbation requiring emergency room treatment within 4 weeks or hospitalisation within 8 weeks of Visit 1.
15. Any use of oral/parenteral corticosteroid within 8 weeks of Visit 1.
16. Surgery to the lower respiratory tract.
17. Hypersensitivity to Ectoin® or any of the other ingredients

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 204 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Morning Peak Expiratory Flow | Baseline (week 1) upto week 4
  Change in mPEF during the treatment period from baseline will be analysed using a model for repeated measurements (MMRM) with time (week), mPEF baseline value and age class (<12 and ≥12 years) as fixed factors and patient as a random effect.
  The morning PEF is to be measured in the morning upon awakening before taking any asthma controller/rescue medication.
  The PEF is defined as the maximum speed of expiration as measured with the Smart Peakflow (best of 3 measurements). The baseline measurement is represented by the mean of the 7 daily values recorded during the run-in period (week 1) and the end-of-treatment measurement is the mean of morning PEF during week 4 (at least 7 days, V3)

SECONDARY OUTCOMES:
Change in Evening Peak Expiratory Flow | Baseline (week 1) to week 2, week 3 and week 4
  Change in weekly mean evening peak expiratory flow (PEF). The evening PEF is to be measured in the evening at bedtime.
Change in Morning/Evening Peak Expiratory Flow | Week 4 to week 5
  Change in weekly mean evening peak expiratory flow (PEF). The evening PEF is to be measured in the evening at bedtime.
Change Morning PEF | Baseline (week 1) to each treatment week (week 2 and week3)
  Change in weekly mean morning peak expiratory flow (PEF). The morning PEF is to be measured in the morning upon awakening before taking any asthma controller/rescue medication.
Rescue medication | Baseline (week 1) upto week 4
  Evolution of the mean number of days with rescue medication
Rescue medication | Week 5
  Evolution of the mean number of days with rescue medication follow-up.
FeNO (fractional exhaled nitric oxide) assessment | Baseline (week 1) upto week 4
  Change of fractional exhaled nitric oxide for a sub-group of patients performed on-site over study visit at selected study sites.
FeNO (fractional exhaled nitric oxide) assessment | Week 4 to week 5
  Change of fractional exhaled nitric oxide for a sub-group of patients performed on-site over study visit at selected study sites follow-up.
Quality of life questionnaire PAQLQ or AQLQ+12 | Week 2 upto week 5
  Change of quality of life assessed by the change of Paediatric Asthma Quality of Life Questionnaire score for children up to 12 years (PAQLQ) and by change of the Asthma Quality of Life Questionnaire for patients 12-year-old and older (AQLQ+12) score for adolescent and adult patients.
Change in Asthma control questionnaire (ACQ-7) | Baseline (week 1) upto week 4
  Change of asthma control questionnaire (ACQ-7) Mean scores of <= 0.75 indicate well-controlled asthma, scores between 0.76 and less than (<) 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma).
Change in Asthma control questionnaire (ACQ-7) | Week 4 to week 5
  Change of asthma control questionnaire (ACQ-7) follow-up Mean scores of <= 0.75 indicate well-controlled asthma, scores between 0.76 and less than (<) 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma).

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej EMERYK, MD, PhD, Principal Investigator — Alergotest, Lublin, Poland
Locations (5):
- Poland (5):
  - Site 5, Bialystok
  - Site 1, Lublin
  - Site 4, Poznan
  - Site 2, Rzeszów
  - Site 3, Warsaw

IPD SHARING:
Plan to Share IPD: No